CLINICAL TRIAL: NCT05589246
Title: Regional Analgesia in Combination With Intraoperative Cryoanalgesia Are the Essential Parts of Enhanced Recovery Protocol in the Minimally Invasive Modyfied Nuss Procedure of Children With Funnel Chest Deformation
Brief Title: Regional Analgesia in Combination With Cryoanalgesia to Prevent Acute Pain Following Nuss Procedure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Jowita Biernawska, Principal Investigator, Pomeranian Medical University Szczecin
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: PomeranianMU-KRIO
Record Dates: First submitted 2022-10-08; First posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Acute Pain; Regional Anesthesia
Keywords: nuss procedure
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): intraoperative cryoanalgesia of intercostal nerves with multimodal analgesia
- intervention (Experimental): regional analgesia (ESP block) with intraoperative cryoanalgesia of intercostal nerves and multimodal analgesia
  Interventions: Device: regional analgesia with cryolesia

INTERVENTIONS:
Device: regional analgesia with cryolesia — The regional analgesia (erector spine plane block) will be added to intraoperative cryolesia of intercostal nerves
  Arms: intervention

SUMMARY:
Funnel chest deformation is a painful procedure, which requires high doses and long time used of opioids. It makes difficult introduction of ERAS protocol. Intraoperative cryolesia of intercostal nerves serves great relief of pain after this procedures. However ablation of the nerves needs 12-24 hours to achieve effects. During this time the high doses of opioids are needed. It causes side effects (sedation makes rehabilitation difficult). On the other hand, percutaneus cryoablation performed 12-24 hours before Nuss procedure needs repeated general anaesthesia. The investigators hypothesed that regional analgesia (erector spine plain block) performed just before intraopertive cryolesia may cover time to full cryolesia effect.

DETAILED DESCRIPTION:
Severe pain in the post-Nuss procedure needs the use of many analgesic drugs, including opioids. It may cause adverse side effects and difficulties with rehabilitation. Moreover, it increases the risk of complications and prolonged hospitalisation. Cryoanalgesia as a part of multimodal analgesia offers better analgesia than single regional techiques with drugs and fasilitate introduction of the enhanced recovery after surgery (ERAS) protocol. However ablation of the nerves needs 12-24 hours to achieve effects. Regional analgesia (erector spine plain block) performed just before intraopertive cryolesia may cover time to full cryolesia effect.

This Before - After Study is a single institution pilot study designed to compare intraoperative cryolesia alone (control group) with the intervention group (cryolesia and bilateral erector spine plane block). It is designed for better management of acute pain in the pediatric population diagnosed with funnel-chest and treated using the modyfied Nuss method. Control group received standard care with cryolesia using the Cryo-S Painless device (Metrum - Cryoflex Polska Limited) and multimodal analgesia according the current guidelines. The intervention group received all of the above and regional analgesia (erector spine plain block, ESP block).

The aims of the study were the assessment the effectiveness of ESP block before full action of intraoperative cryoanalgesia as a method of acute pain control, safety of the method.

The results were compared in terms of demographics, pain levels, side effects of the pain relief medications in the postoperative period and lenght of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing pectus excavatum repair with modyfied minimal invasive thoracoscopic NUSS technique
* aged 10 years or above 10 up to 18
* informed consent signed for cryoanalgesia informed consent signed for regional analgesia

Exclusion Criteria:

* Age of 9 years or below
* Refuse to receive cryoanalgesia or regional analgesia as primary pain relief
* Any contraindication to cryoanalgesia
* Difficult follow-up for geographical reasons and/or impossibility by the patient to understand how to perform self-measurements

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The worse pain | within first 24 hours after operation
  Maximal pain within first 24 hours after operation, Numeric pain score. Range from 0 to 10.

SECONDARY OUTCOMES:
LAST (Local anesthetic systemic toxicity) | within first 24 hours after operation
  No score exists. Assesment of clinical features: sensory and visual changes, muscular activation, seizure activity, new rhythm disturbances.

CONTACTS AND LOCATIONS:
Overall Officials: Jowita Biernawska, MD PhD, Principal Investigator — Pomeranian Medical Universitet Szczecin
Locations (1):
- Pomeranian Medical University, Szczecin, Poland

IPD SHARING:
Plan to Share IPD: Undecided
after contact with the principal investigator